CLINICAL TRIAL: NCT06143163
Title: Clinical Outcome of Treatment of Ulcerative Colitis in Adult.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kholoud Mohamed Hassan, Dr kholoud Mohamed Hassan, Assiut University
Other Study IDs: Treatment of UC
Record Dates: First submitted 2023-11-05; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. characterize the response to current medical therapy in adult with ulcerative colitis .
2. Detect prognostic factors of response of biological therapy in adult with ulcerative colitis

DETAILED DESCRIPTION:
Ulcerative colitis is an idiopathic inflammatory condition of the colon which results in diffuse friability and superficial erosions on the colonic wall associated with bleeding. It is the most common form of inflammatory bowel disease worldwide. It characteristically involves inflammation restricted to the mucosa and submucosa of the colon. Typically, the disease starts in the rectum and extends proximally in a continuous manner. In the United States, the disease accounts for a quarter-million provider visits annually, and medical costs directly related to the disease are estimated to exceed four billion dollars annually.Ulcerative has no cure and is a lifelong disorder with a significant impact on both physical and mental health. The specific cause of inflammatory bowel disease is not known. There seems to be a primary genetic component since the most important independent risk factor is a family history of the disease (8% to 14% of patients). A first-degree relative of a patient with ulcerative colitis has a four times higher risk of developing the disease. Although there is little evidence to support this, it has been postulated that alterations in the composition of the gut microbiota and defects in mucosal immunity could lead to ulcerative colitis. Autoimmunity may also play an important role in the etiology of ulcerative colitis.Diagnosis of ulcerative colitis is made clinically with supportive findings on endoscopy, biopsy, and by negative stool examination for infectious causes. Because colonic infection can produce clinical findings indistinguishable from idiopathic ulcerative colitis, microbiologic studies for bacterial infection and parasitic infestation should be included in the initial evaluation.Treatment choice for patients with ulcerative colitis is based on both the extent of the disease and the severity. The prognosis during the first decade after diagnosis is often generally good, and most patients go into remission. Rectal application of medical therapy, via suppository or enema, is usually appropriate for isolated distal disease (proctitis); however, a rectal application is usually used in combination with systemic therapy to help target the distal colon and therefore decrease tenesmus.Ulcerative colitis has no cure and despite treatment, many continue to have increased bouts of stool frequency. An increase in mortality is usually seen in elderly patients, those with complications like infection, shock, anemia, and those who require repeated surgical interventions. Data show that when the disease involves the muscularis propria, it can lead to bowel dysmotility, necrosis, and gangrene. A certain number of patients also develop toxic megacolon with poor outcomes. It is estimated that about 5% of patients will develop colorectal cancer over time. The risk of colon cancer is higher in patients with pancolitis and in patients whose disease started before the age of 15. Overall, the quality of life in patients with ulcerative colitis is poor.

ELIGIBILITY:
Inclusion Criteria:

* All Patients above age of 18 years old previously diagnosed by colonscopy and biobsy with ulcerative colitis attending IBD clinic El-Raghy liver Hospital

Exclusion Criteria:

1. patients younger than 18 years old .
2. patients known to have chronic liver disease.
3. patient known to have renal disease.
4. Patients diagnosed with cardiac disease.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. diagnosed by colonscopy and biobsy with ulcerative colitis .
  2. must be above 18yrs.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2024-12-29 (Estimated); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
- Characterize the response to current medical therapy in adult with Ulcerative colitis | Baseline
  The clinical course of the disease Will be assessed after 3 months of treatment according to guidelines as follow
  1. clinical assessment as regard symptoms as rectal bleeding, diarrhea, abdominal pain, stool frequency guided by mayo score.
  2. laboratory assessment including: ESR,CRP,CBC,fecalcalprotectin.
  3. Endoscopic evaluation regarding the mayo score.
  4. Histopathological assessment to evaluate the stage of activity of the disease.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gisbert JP, Chaparro M. Clinical Usefulness of Proteomics in Inflammatory Bowel Disease: A Comprehensive Review. J Crohns Colitis. 2019 Mar 26;13(3):374-384. doi: 10.1093/ecco-jcc/jjy158. PMID 30307487
- [Background] Jackson B, De Cruz P. Algorithms to facilitate shared decision-making for the management of mild-to-moderate ulcerative colitis. Expert Rev Gastroenterol Hepatol. 2018 Nov;12(11):1079-1100. doi: 10.1080/17474124.2018.1530109. Epub 2018 Oct 17. PMID 30284911
- [Background] Spiceland CM, Lodhia N. Endoscopy in inflammatory bowel disease: Role in diagnosis, management, and treatment. World J Gastroenterol. 2018 Sep 21;24(35):4014-4020. doi: 10.3748/wjg.v24.i35.4014. PMID 30254405
- [Background] Ashton JJ, Ennis S, Beattie RM. Early-onset paediatric inflammatory bowel disease. Lancet Child Adolesc Health. 2017 Oct;1(2):147-158. doi: 10.1016/S2352-4642(17)30017-2. Epub 2017 Aug 7. PMID 30169204
- [Background] Guardiola J, Lobaton T, Cerrillo E, Ferreiro-Iglesias R, Gisbert JP, Domenech E, Chaparro M, Esteve M, Rodriguez-Moranta F; en representacion de GETECCU. Recommendations of the Spanish Working Group on Crohn's Disease and Ulcerative Colitis (GETECCU) on the utility of the determination of faecal calprotectin in inflammatory bowel disease. Gastroenterol Hepatol. 2018 Oct;41(8):514-529. doi: 10.1016/j.gastrohep.2018.05.029. Epub 2018 Jul 4. English, Spanish. PMID 30293556
- [Background] Lee JS, Kim ES, Moon W. Chronological Review of Endoscopic Indices in Inflammatory Bowel Disease. Clin Endosc. 2019 Mar;52(2):129-136. doi: 10.5946/ce.2018.042. Epub 2018 Aug 21. PMID 30130840
- [Background] Danese S, Banerjee R, Cummings JF, Dotan I, Kotze PG, Leong RWL, Paridaens K, Peyrin-Biroulet L, Scott G, Assche GV, Wehkamp J, Yamamoto-Furusho JK. Consensus recommendations for patient-centered therapy in mild-to-moderate ulcerative colitis: the i Support Therapy-Access to Rapid Treatment (iSTART) approach. Intest Res. 2018 Oct;16(4):522-528. doi: 10.5217/ir.2018.00073. Epub 2018 Oct 16. PMID 30321913
- [Background] Rodriguez-Lago I, Ferreiro-Iglesias R, Nos P, Gisbert JP; en representacion del Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (GETECCU). Management of acute severe ulcerative colitis in Spain: A nationwide clinical practice survey. Gastroenterol Hepatol. 2019 Feb;42(2):90-101. doi: 10.1016/j.gastrohep.2018.09.002. Epub 2018 Oct 4. English, Spanish. PMID 30293913
- [Background] Borman ZA, Cote-Daigneault J, Colombel JF. The risk for opportunistic infections in inflammatory bowel disease with biologics: an update. Expert Rev Gastroenterol Hepatol. 2018 Nov;12(11):1101-1108. doi: 10.1080/17474124.2018.1530983. Epub 2018 Oct 10. PMID 30277409
- [Background] Drews JD, Onwuka EA, Fisher JG, Huntington JT, Dutkiewicz M, Nogalska A, Nwomeh BC. Complications after proctocolectomy and ileal pouch-anal anastomosis in pediatric patients: A systematic review. J Pediatr Surg. 2019 Jul;54(7):1331-1339. doi: 10.1016/j.jpedsurg.2018.08.047. Epub 2018 Sep 19. PMID 30291026